CLINICAL TRIAL: NCT04835506
Title: Proactive Infliximab Optimization Using a Pharmacokinetic Dashboard Versus Standard of Care in Patients With Inflammatory Bowel Disease: The OPTIMIZE Trial
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Adam Cheifetz, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000391
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- proactive infliximab optimization (Experimental): proactive infliximab optimization using a pharmacokinetic dashboard
  Interventions: Drug: Infliximab
- standard of care infliximab dosing (Experimental): standard of care infliximab dosing
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — infliximab

SUMMARY:
The OPTIMIZE Trial compares whether iDose dashboard-driven infliximab dosing (iDose-driven dosing) is more effective and safer than standard infliximab dosing for inducing and maintaining disease remission in inflammatory bowel disease.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), namely Crohn's disease (CD) and ulcerative colitis (UC) are life-long chronic diseases characterized by transmural inflammation of the intestine. CD and UC are global diseases in the 21st century with increasing incidence in newly industrialized countries. One of the most effective therapies to treat patients with moderate to severe disease is the antitumor necrosis factor (TNF) agent infliximab (IFX) either as monotherapy or as a combination therapy with an immunomodulator (IMM), such as azathioprine or methotrexate (MTX).

Although more effective, combination therapy is associated with more serious adverse events, such as serious opportunistic infections and cancers, as well as potential treatment adherence issues. Consequently, many patients and physicians choose to use IFX alone as safety is often prioritized over efficacy. Unfortunately, up to 30% of patients do not respond to induction therapy, and up to 50% of initial responders lose response over time. It is only if patients lose response that physicians check blood IFX concentrations (i.e., reactive therapeutic drug monitoring [TDM]), or empirically increase IFX dose. Reactive TDM helps to explain and better manage these patients with lack or loss of response to IFX. In many cases, the lack or LOR is due to low drug concentrations with or without development of antibodies to IFX (ATI). Unfortunately, reactive TDM or empiric dose escalation is often too late for patients who do not either respond to IFX induction therapy or lose response during maintenance. This reactive approach results in many patients losing IFX as a therapeutic option.

Preliminary data show that proactive IFX optimization to achieve a threshold drug concentration during maintenance therapy (even if the patient is asymptomatic) compared to empiric dose escalation and/or reactive TDM is associated with better long-term outcomes including longer drug persistence, reduced risk of relapse, and fewer hospitalizations and surgeries. IFX dosing by weight only (i.e., mg/kg) may not be adequate for many patients as interindividual variability in drug clearance and other factors affecting IFX concentrations and PK are often not accounted for. Dosing calculators take into account all of these individual factors and improve the precision of dosing towards better personalized medicine. These systems have already been validated, and personalized dosing has shown clinical benefit in patients with IBD.

This is a randomized, controlled, multicenter, open-label study that plans to enroll 196 participants with inflammatory bowel disease. All eligible participants will be randomly assigned in a 1:1 ratio to receive either IFX monotherapy with proactive TDM or SOC IFX therapy, with or without concomitant IMM therapy, and empiric dose optimization or reactive TDM, at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Males or nonpregnant, nonlactating females aged 16 to 80 years inclusive.
2. Diagnosis of IBD prior to screening using standard endoscopic, histologic, or radiologic criteria. Participants with patchy colonic inflammation initially diagnosed as indeterminate colitis would meet inclusion criteria, if the investigator feels that the findings are consistent with CD or UC. Enrollment of participants with UC will be capped at 49% of the planned study population (maximum 61 participants).
3. Moderately to severely active IBD, defined by a total CDAI score between 220 and 450 points for CD or a partial Mayo Score (PMS) > 4 for UC (including a rectal bleeding subscore [RBS] ≥ 1), and at least 1 of the following:

   1. Elevated CRP (> upper limit of normal)
   2. Elevated FC (> 250 μg/g)
   3. SES-CD > 6 (SES-CD > 3 for isolated ileal disease) for CD only and a Mayo endoscopic subscore (MES) ≥ 2 for UC only.
4. Physician intends to prescribe IFX as part of the usual care of the subject.
5. No previous use of IFX prior to enrolment in the current study, unless the participant received 1 prior dose of IFX (within 2.5 weeks of enrolment) and met all eligibility criteria at the time of starting IFX and IFX was administered according to the requirements outlined in this protocol
6. Able to participate fully in all aspects of this clinical trial.
7. Written informed consent must be obtained and documented.

Exclusion Criteria:

1. Participants with any of the following IBD-related complications:

   1. Abdominal or pelvic abscess, including perianal
   2. Presence of stoma, ileal pouch-anal anastomosis, or ostomy
   3. Isolated perianal disease
   4. Obstructive disease, such as obstructive stricture
   5. Short gut syndrome
   6. Toxic megacolon or any other complications that might require surgery, or any other manifestation that precludes or confounds the assessment of disease activity (CDAI or SES-CD for CD or PMS, PRO2, or MES for UC)
   7. Total colectomy.
2. History or current diagnosis of ulcerative proctitis (UC extending < 15 cm from the anal verge), acute severe (fulminant) UC, hospitalised IV steroid-refractory UC, indeterminate colitis, microscopic colitis, ischemic colitis, colonic mucosal dysplasia, or untreated bile acid malabsorption.
3. Current bacterial or parasitic pathogenic enteric infection, according to SOC assessments, including: Clostridioides difficile; tuberculosis; known infection with hepatitis B or C virus; known infection with HIV; sepsis; abscesses. History of the following: opportunistic infection within 6 months prior to screening; any infection requiring antimicrobial therapy within 2 weeks prior to screening; more than 1 episode of herpes zoster or any episode of disseminated zoster; any other infection requiring hospitalization or intravenous antimicrobial therapy within 4 weeks prior to screening.
4. Has any malignancy or lymphoproliferative disorder other than nonmelanoma cutaneous malignancies or cervical carcinoma in situ that has been treated with no evidence of recurrence within the last 5 years.
5. Known primary or secondary immunodeficiency.
6. PNR to adalimumab, defined as no objective evidence of clinical benefit after 14 weeks of therapy.
7. Subjects with failure to a prior biologic, defined as PNR or SLR, will be excluded when a maximum of 40% of the planned enrollment (approximately 78 subjects) have failure to prior biologic exposure.
8. Concomitant use of oral corticosteroid therapy exceeding prednisone 40 mg/day, budesonide 9 mg/day, or equivalent, unless a tapering schedule is initiated with a plan to be off CS by Week 14
9. Presence of any medical condition or use of any medication that is a contraindication for IFX use, as outlined on the product label.
10. A concurrent clinically significant, serious, unstable, or uncontrolled underlying cardiovascular, pulmonary, hepatic, renal, GI, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, might confound the study results, pose additional risk to the subject, or interfere with the subject's ability to participate fully in the study.
11. Pregnant or lactating women, to be excluded based on the physician's usual practice for determining pregnancy or lactation status.
12. Known intolerance or hypersensitivity to IFX or other murine proteins.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical remission | 52 weeks
  Proportion of subjects with sustained corticosteroid-free (no CS use from Week 14 through 52) clinical remission (CD: CDAI <150 at Weeks 14, 26, 52; UC: PRO2 ≤ 1 with an RBS = 0) and no disease worsening

SECONDARY OUTCOMES:
clinical remission | 52 weeks
  Proportion of subjects in CS-free clinical remission (CD: CDAI < 150; UC: PRO2 ≤ 1 with an RBS = 0) and no use of CS within previous 6 months)
deep remission | 52 weeks
  Proportion of subjects in deep remission (CD: CDAI < 150 and SES-CD ≤ 4, with no individual subscore > 1; UC: PRO2 ≤ 1 with an RBS = 0 and MES ≤ 1)
composite biological and endoscopic remission | 52 weeks
  Proportion of subjects with a composite biological (hs-CRP < 10 mg/L) and endoscopic remission (CD: SES-CD ≤ 4; UC: MES ≤ 1)
sustained CS-free clinical remission | 52 weeks
  Proportion of subjects with sustained CS-free clinical remission (CD: CDAI < 150; UC: PRO2 ≤ 1 with an RBS = 0) and no CS use or need for rescue therapy from Week 14 through Week 52)
primary non-responders | 14 weeks
  Proportion of subjects who are primary nonresponders (≤ 70-point decrease in CDAI score or lack of a ≥ 1-point and 30% reduction from baseline in PRO2 and a ≥ 1-point reduction in RBS or an absolute RBS ≤ 1 for UC and at least one of: hs-CRP ≥10 mg/L, FC > 250 μg/g, or SES-CD > 4 or MES > 1 for UC, or disease worsening prior to Week 14)
biological remission | 52 weeks
  Proportion of subjects with sustained biological remission (hs-CRP <10 mg/L)
endoscopic remission | 52 weeks
  Proportion of subjects with endoscopic remission (SES-CD ≤ 4, with no individual subscore > 1 for CD or MES ≤ 1 for UC)
hs-CRP normalization | 52 weeks
  Proportion of subjects with normalization of hs-CRP (decrease from ≥ 10 at baseline to < 10 mg/L)
hs-CRP change from baseline | week 14, week 26, and week 52
  Hs-CRP change from baseline
endoscopic response | 52 weeks
  Proportion of subjects with an endoscopic response (CD: ≥ 50% decrease from baseline SES-CD score; UC: ≥ 1-point decrease in MES)
fecal calprotectin | 52 weeks
  Proportion of subjects with normalization of fecal calprotectin (decrease from >250 µg/g at baseline to ≤ 250 µg/g)
fecal calprotectin change | 52 weeks
  fecal calprotectin change from baseline

CONTACTS AND LOCATIONS:
Locations (25):
- United States (23):
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Rockford GI, Rockford, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Atrium Health Center for Digestive Health, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - LifeSpan Brown University, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - London Health Sciences Centre - Children's Hospital, London
  - McGill University Health Centre (MUHC) Montreal General Hospital, Montreal

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data and trial-level data will be available on reasonable request. This data will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing agreement
Time Frame: After completion and publication of primary study.
Access Criteria: This data will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing agreement

REFERENCES:
- [Derived] Papamichael K, Jairath V, Zou G, Cohen B, Ritter T, Sands B, Siegel C, Valentine J, Smith M, Vande Casteele N, Dubinsky M, Cheifetz A. Proactive infliximab optimisation using a pharmacokinetic dashboard versus standard of care in patients with Crohn's disease: study protocol for a randomised, controlled, multicentre, open-label study (the OPTIMIZE trial). BMJ Open. 2022 Apr 1;12(4):e057656. doi: 10.1136/bmjopen-2021-057656. PMID 35365535